CLINICAL TRIAL: NCT05330598
Title: Evaluation of the Safety and Clinical Performance of the Connected Catheter - Wireless Urinary Prosthesis for Management of Chronic Urinary Retention
Brief Title: Evaluation of the Safety and Clinical Performance of the Connected Catheter Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Spinal Singularity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0003
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Urinary Retention; Chronic
Keywords: Intermittent Catheter; Intermittent catheterization; Urinary retention; Impaired bladder
MeSH Terms: conditions — Urinary Retention; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Connected Catheter Users (Experimental): Device: Connected Urinary Catheter Patients will use the Connected Catheter to empty the bladder during the course of treatment.
  Interventions: Device: Connected Catheter

INTERVENTIONS:
Device: Connected Catheter — The Connected Catheter System is a replaceable wireless urinary prosthesis that is indicated for bladder emptying in male patients who have impaired bladder emptying due to chronic Urinary Retention. The Connected Catheter resides fully internally in the male lower urinary tract (urethra and bladder neck) and remains in place for up to 7 days before removal.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Connected Catheter in males with chronic Urinary Retention, both in a clinical setting and an extended period of home use.

The Connected Catheter is a fully internal, urethral indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization. It is a sterile, extended-use device that resides fully internally to the male lower urinary tract for an intended use life of up to 7 days per catheter.

DETAILED DESCRIPTION:
UroDev Medical has developed the Connected Catheter System to address several drawbacks of urinary catheters. The Connected Catheter is fully internal, indwelling urinary prosthesis designed for improved bladder management in males with urinary retention disorders requiring catheterization. Each subject will use the Connected Catheter for up to 4 weeks including weekly device exchange appointments. Additionally, weekly follow-up will occur for 14 days following the final appointment after the subject discontinues use of study device and reverts to his original catheter.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males > 22 years old diagnosed with chronic Urinary Retention 2. Must be clinically suitable and capable of safely managing bladder using an intermittent voiding or indwelling catheter strategy:

  1. Must have stable urinary management history as determined by the Principal Investigator OR
  2. Must have urodynamic profile suitable for the Connected Catheter (including bladder capacity ≥ 200mL without uninhibited bladder contractions) 3. Subject's lower urinary tract anatomy must fall within the ranges serviceable by the Connected Catheter device, as specified in the Investigational Device Instructions For Use.

Exclusion Criteria:

* 1. Active symptomatic urinary tract infection, as defined in this clinical investigation plan (CIP)/protocol (subjects may receive the device after their UTI has been treated) 2. Significant risk profile or recent history of urethral stricture (e.g., stricture within past 90 days) 3. Significant risk profile or recent history of clinically significant (uncontrolled) autonomic dysreflexia 4. Significant intermittent urinary incontinence (between catheterizations) 5. Uninhibited bladder contractions and/or Vesicoureteral reflux that is not reliably controlled with medication or alternate therapy (e.g., Botox injection)

  1. Active symptomatic urinary tract infection, as defined in this clinical investigation plan (CIP)/protocol (subjects may receive the device after their UTI has been treated)
  2. Significant risk profile or recent history of urethral stricture (e.g., stricture within past 90 days)
  3. Significant risk profile or recent history of clinically significant (uncontrolled) autonomic dysreflexia
  4. Significant intermittent urinary incontinence (between catheterizations)
  5. Uninhibited bladder contractions and/or Vesicoureteral reflux that is not reliably controlled with medication or alternate therapy (e.g., Botox injection)
  6. Pre-existing urinary pathologies and/or morphological abnormalities of the lower urinary tract or bladder (assessed during in-depth medical screening, including cystoscopy and urine analysis)

     1. Urinary tract inflammation or neoplasm
     2. Urinary fistula
     3. Bladder diverticulum (outpouching) > 5cm in size
     4. Chronic pyelonephritis (secondary to upper urinary tract infection(s) within past 6 months)
     5. Impaired kidney function or renal failure
     6. Active gross hematuria
     7. Active urethritis
     8. Bladder stones
  7. Dependence on an electro-magnetic medical implant (e.g., cardiac pacemaker or implanted drug pump) or external device
  8. Any unsuitable comorbidities as determined by the Principal Investigator or complications related to use of certain medications
  9. Any physical or cognitive impairments that diminish the subject's ability to follow directions or otherwise safely use the Connected Catheter System
  10. Catheter Assessment Tool screening yields unacceptable results
  11. Vulnerable population such as inmates or developmentally delayed adults

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The connected catheter is designed for male use.
Enrollment: 26 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Successful Bladder Emptying Using Connected Catheter | 4 weeks
  PVR Responder Rate, defined as either:
  * Less than or equal to 50mL OR
  * Equal to or less than their baseline PVR when using SOC catheters
  The subject responder rate, R, is estimated as the proportion of subjects who are classified as responders.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rancho Research Institute, Downey, California
  - West Coast Urology, 575 E. Hardy St., Suite 215, Inglewood, California
  - Tri Valley Urology, 25495 Medical Center Dr., Suite 204, Murrieta, California
  - UCSD, San Diego, California
  - Medstar National Rehabilitation Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No